CLINICAL TRIAL: NCT02794441
Title: Oral Dexamethasone for the Treatment of Acute Migraine Recurrence in Pediatric Patients Presenting to the Emergency Department With Migraine: A Pilot Randomized Controlled Trial
Brief Title: Oral Dexamethasone for the Treatment of Acute Migraine Recurrence in the Pediatric Emergency Department
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Roger Zemek, Scientist, CHEO Research Institute; Director, CHEO Research Institute Clinical Research Unit; Emergency Physician, CHEO, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20150453
Record Dates: First submitted 2016-05-25; First posted 2016-06-09 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone 0.6mg/kg (maximum 15mg) PO x 1 dose
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator): Matched oral solution in same volume per kg as dexamethasone
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 0.6mg/kg (maximum 15mg) PO x 1 dose
  Arms: Dexamethasone
Other: Placebo — Matched oral solution
  Arms: Placebo

SUMMARY:
Migraine recurrence is common amongst pediatric patients being discharged from the emergency department after treatment for migraine. Despite the commonality of migraine recurrence within the week following discharge, no known effective therapies are available in the pediatric population, though dexamethasone has been established as efficacious in the adult migraine population. The proposed study will randomly assign children and adolescents visiting the emergency department (ED) for migraine to receive either one dose of oral dexamethasone or oral placebo. Twenty patients will be recruited to this randomized, double-blind, pilot trial over a 6 month period, and the aim of the study will be to determine the feasibility and acceptability of the protocol.

DETAILED DESCRIPTION:
Migraine is common in the pediatric emergency department. Unfortunately, somewhere between one third and two thirds of children and adolescents will have recurrence of their migraine within a week of discharge from the emergency department. Although there is strong evidence from adult studies that dexamethasone can prevent migraine recurrence, there is no evidence on how to prevent recurrence in children and adolescents. The proposed study will randomly assign children and adolescents visiting the Children's Hospital of Eastern Ontario (CHEO) emergency department (ED) for migraine to receive either one dose of oral dexamethasone or oral placebo. Twenty patients will be recruited to this randomized, double-blind, pilot trial over a 6 month period, and the aim of the study will be to determine the feasibility and acceptability of the protocol.

Patients will be recruited from the CHEO ED. Research volunteers will screen patients with a triage diagnosis of 'headache', 'migraine' or a related triage diagnosis for eligibility. Patients who meet eligibility criteria will be approached by a research assistant who will initiate the consent process. Informed consent will be sought through both verbal explanation and in written form, from participants 14 years and over and from the parent(s) or guardian(s). For participants under the age of 14 years, verbal and written assent will be sought.

Consenting participants will be randomized to receive one dose of oral dexamethasone 0.6mg/kg to a maximum of 15mg or one dose of oral matched placebo. Randomization will be stratified by baseline migraine duration: 1) less than 2 hours, 2) 2 hours to less than 24 hours and 3) 24 hours and greater. A list of randomization codes will be generated over the computer by a biostatistician and randomization will occur in blocks of four. Research personnel will not have access to the randomization code list with group assignments. Only the research pharmacists will have access to the list.

The research assistants will collect outcome data from the participants and store it into Research Electronic Data Capture (REDCaP), a secure, encrypted web-based platform. Participants will have the option of completing follow-up via email questionnaires or over the telephone. Follow-up will take place 48 hours and 7 days after discharge. The purpose of follow-up will be to assess whether or not participants had recurrence of their migraine, and to collect other follow-up outcome data and safety data. The research assistants, participants, research personnel and clinical personnel will all be blinded to group assignment. Only the research pharmacists, who will not interact with anyone in the study directly, will have access to group assignment information.

Data analyses will be carried out for exploratory purposes, and the groups (dexamethasone vs. placebo) will be compared with regards to: baseline data, 48 hour migraine recurrence rates, 7 day migraine recurrence rates, the proportion of participants achieving pain freedom at 2 hours and maintaining it at 48 hours, patient satisfaction data and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 8 and 18 years (ie. > 8.0 years and < 18.0 years)
2. Diagnosed with migraine according to a modified version of International Classification of Headache Disorders 3rd edition (ICHD-3, beta version) where criterion A (ie. minimum of 5 prior episodes meeting criteria B-D) has been removed to increase sensitivity of diagnosis in the emergency department setting

Exclusion Criteria:

1. Received a dose of a steroid medication in the past 7 days
2. Known allergy to dexamethasone
3. Immunosuppressed
4. Cushing's syndrome
5. Known diabetes mellitus
6. Known peptic or duodenal ulcer or other major gastrointestinal illness (ex. ulcerative colitis)
7. Known myasthenia gravis
8. Glaucoma
9. Febrile at triage
10. History of head trauma in the past 7 days
11. Presence of any known active infection (eg. on antibiotics or antivirals, diagnosed with active infection in the ED, etc)
12. Current secondary headache (as per the treating physician's clinical impression)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2016-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Zemek, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tfelt-Hansen P, Pascual J, Ramadan N, Dahlof C, D'Amico D, Diener HC, Hansen JM, Lanteri-Minet M, Loder E, McCrory D, Plancade S, Schwedt T; International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine: third edition. A guide for investigators. Cephalalgia. 2012 Jan;32(1):6-38. doi: 10.1177/0333102411417901. No abstract available. PMID 22384463
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between December 2016 and June 2017 from the ED at the Children's Hospital of Eastern Ontario, a tertiary care academic pediatric hospital located in Ottawa, Ontario, Canada.
Period: Overall Study
Arm/Group | Dexamethasone | Placebo
Started | 7 | 5
Completed | 6 | 5
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: One participant in the dexamethasone group withdrew from the study prior to receiving the study intervention and is not included in the analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.6 (3.4) | 13.6 (0.9) | 13.0 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 1 | 3 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 5 | 11
CTAS Score [Count of Participants; unit: Participants]
  Resuscitation | 0 | 0 | 0
  Emergent | 0 | 0 | 0
  Urgent | 6 | 4 | 10
  Semi-Urgent | 0 | 1 | 1
  Non-Urgent | 0 | 0 | 0
Baseline Pain Intensity [Count of Participants; unit: Participants]
  None | 0 | 0 | 0
  Mild | 0 | 0 | 0
  Moderate | 2 | 1 | 3
  Severe | 4 | 4 | 8
Use of Treatment at Home [Count of Participants; unit: Participants]
  Yes | 4 | 5 | 9
  No | 2 | 0 | 2
Migraine Type [Count of Participants; unit: Participants]
  Migraine with aura | 4 | 5 | 9
  Migraine without aura | 3 | 0 | 3
Headache Frequency (Monthly Frequency in Past 3 Months) [Mean (Standard Deviation); unit: Headaches] | 12.6 (12.9) | 7.2 (12.8) | 10.3 (12.6)
How Long Participant Has Had Migraines [Mean (Standard Deviation); unit: years] | 5.1 (9.9) | 2.0 (1.6) | 3.6 (6.8)
PedMIDAS Score [Mean (Standard Deviation); unit: units on a scale] — PedMIDAS: The Pediatric Migraine Disability Assessment Scale measures migraine-specific disability in children and adolescents. The minimum score is 0 and the maximum score is 240. Lower scores indicate less migraine-specific disability and higher scores indicate higher migraine-specific disability. Scores ranging from 0-10 indicate grade I (little-no disability), scores from 11-30 indicate grade II (mild disability), scores from 31-50 indicate grade III (moderate disability) and scores over 50 indicate grade IV (severe disability).
  units on a scale | 58.7 (108.5) | 16.2 (17.8) | 41 (83.8)

OUTCOME MEASURES:

1. Primary Outcome: Headache Recurrence at 48 Hours
Description: The primary outcome will be headache recurrence 48 hours after discharge from the ED. Headache recurrence will be defined as: for patients who were pain-free at ED discharge (ie. pain intensity of 0), any return of head pain (ie. pain intensity of 1 or greater) will be coded as a recurrence, and for patients who had persistent head pain at discharge, an increase in head pain since ED discharge will be coded as recurrence as well (ie. an increase in their score on the 4-point scale as compared to their score at ED discharge).
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 1 | 1

2. Secondary Outcome: Pain Intensity
Description: Pain intensity will be measured on a 4 point rating scale as recommended by the International Headache Society guidelines: a) 0=none, b) 1=mild, c) 2= moderate, d) 4=severe. It will be assessed at 2 hours post-baseline, or at the time of ED discharge if prior to 2 hours and at the time of ED discharge where this exceeds 2 hours post-intervention. Because all participants were discharged prior to 2 hours, we report the pain intensity at the time of ED discharge.
Time Frame: Baseline, 2 hours post-intervention (or at the time of ED discharge if prior to 2 hours) and at the time of discharge from the Emergency Department (ED) if post-treatment ED duration extends beyond 2 hours (expected median duration = 3 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  None | 2 | 1
  Mild | 2 | 2
  Moderate | 2 | 2
  Severe | 0 | 0

3. Secondary Outcome: Persistent Pain Freedom
Description: Persistent pain freedom, defined as the proportion of patients in each group who achieved pain freedom at 2 hours (or at the time of ED discharge if prior to 2 hours) and were free of pain without the use of rescue medication at 48 hours, will be assessed
Time Frame: 2 hours post-intervention (or at the time of ED discharge if prior to 2 hours) and 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 1 | 1

4. Secondary Outcome: Patient Satisfaction
Description: Patient satisfaction will be assessed at the time of discharge from the ED and again at follow-up with the following 5-point Likert scale: 5=very satisfied, 4=satisfied, 3=neutral, 2=unsatisfied, 1=very unsatisfied. Here we report patient satisfaction rates at discharge.
Time Frame: At the time of discharge from the ED (expected median duration in the ED post-treatment = 3 hours), at 48 hours and at 7 day follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  At discharge: Satisfied | 6 | 4
  At discharge: Dissatisfied | 0 | 1
  At 48 hour follow-up: Satisfied | 6 | 4
  At 48 hour follow-up: Dissatisfied | 0 | 1
  At 7 day follow-up: Satisfied | 6 | 3
  At 7 day follow-up: Dissatisfied | 0 | 2

5. Secondary Outcome: Headache Recurrence at 7 Day Follow-up
Description: The proportion of patients in each group with recurrence within the 7 days following ED discharge will be assessed.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 0 | 0

6. Secondary Outcome: Revisits Within 7 Days of Discharge From the ED
Description: The number of patients with return ED visits within 7 days of ED discharge will be assessed through chart review.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 6 | 5
Participants | 1 | 0

7. Secondary Outcome: Adverse Events at Discharge
Description: Adverse events will be queried at 2 hours (or at the time of ED discharge if prior to 2 hours), at discharge and in the follow-up questionnaires at 48 hours and 7 days. Reported here are the adverse events at the time of ED discharge. All patients were discharged prior to the 2 hour time point. Adverse events reported at follow-up are reported elsewhere (see below).
Time Frame: 2 hours post-intervention (or at the time of ED discharge if prior to 2 hours), at the time of discharge from the Emergency Department (ED) if post-treatment ED duration extends beyond 2 hours (expected median duration = 3 hours), 48 hours and 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  Adverse events | 0 | 0
  No adverse events | 6 | 5

8. Secondary Outcome: Adverse Events at 48 Hours Post-discharge
Description: Adverse events will be queried at 2 hours (or at the time of ED discharge if prior to 2 hours), at discharge and in the follow-up questionnaires at 48 hours and 7 days. Reported here are the adverse events at the 48 hour follow-up post-discharge.
Time Frame: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  Worsening headache | 1 | 1
  Fever | 0 | 1
  Constipation | 1 | 0
  No adverse events | 4 | 3

9. Secondary Outcome: Adverse Events at 7 Days Post-discharge
Description: Adverse events will be queried at 2 hours (or at the time of ED discharge if prior to 2 hours), at discharge and in the follow-up questionnaires at 48 hours and 7 days. Reported here are the adverse events at the 7 day follow-up post-discharge.
Time Frame: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 6 | 5
Participants
  Paresthesias | 0 | 1
  Headache recurrence | 0 | 1
  No adverse events | 6 | 3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at discharge and for the first 7 days after discharge
Description: The medication (dexamethasone) has potential to cause immunosuppression.
Arm/Group | Dexamethasone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 2/6 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=6) | Placebo (N=5)
Worsening headache (Nervous system disorders) | 1 (1) | 1 (1) — Patients reporting worsening of their headache post-discharge
Paresthesias (Nervous system disorders) | 0 (0) | 1 (1) — Patient reporting transient self-resolving parenthesis of the upper lip
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — Patient reporting 3 days with no bowel movement after discharge. The constipation self-resolved.
Fever (General disorders) | 0 (0) | 1 (1) — One participant had fever post-discharge that resolved

LIMITATIONS AND CAVEATS:
This study was designed as a pilot trial to assess trial protocol feasibility. Statistical hypothesis testing was not conducted on any of the outcome variables because of the small sample size and the inability to draw inferences from this data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT02794441/Prot_SAP_000.pdf